CLINICAL TRIAL: NCT02404350
Title: A Phase III, Randomized, Double-blind, Placebo Controlled Multi-center Study of Subcutaneous Secukinumab (150 mg and 300 mg) in Prefilled Syringe to Demonstrate Efficacy (Including Inhibition of Structural Damage), Safety, and Tolerability up to 2 Years in Subjects With Active Psoriatic Arthritis (FUTURE 5)
Brief Title: Study to Demonstrate the Efficacy (Including Inhibition of Structural Damage), Safety and Tolerability up to 2 Years of Secukinumab in Active Psoriatic Arthritis
Acronym: FUTURE5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2342; 2015-000050-38 (EudraCT Number); 02404350 (Registry Identifier: clinicaltrials.gov)
Record Dates: First submitted 2015-03-16; First posted 2015-03-31 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Arthritis; Psoriatic; Psoriatic Arthropathy; Spondylitis
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis; Spondylitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Secukinumab 150 mg load (Group 1) (Experimental): Secukinumab 150 mg sc injection every week for 4 weeks followed by Secukinumab 150 mg every 4 weeks until week 100
  Beginning at Week 52, for subjects whose signs and symptoms were not fully controlled, and who the investigator believed may improve further with an increase in dose, may have had the secukinumab dose increased to 300mg s.c. every 4 weeks until week 100
  Interventions: Biological: Secukinumab
- Secukinumab 150 mg no load (Group 2) (Experimental): Secukinumab 150 mg sc injection every 4 weeks until week 100
  Beginning at Week 52, for subjects whose signs and symptoms were not fully controlled, and who the investigator believed may improve further with an increase in dose, may have had the secukinumab dose increased to 300mg s.c. every 4 weeks.
  Interventions: Biological: Secukinumab
- Secukinumab 300 mg load (Group 3) (Experimental): Secukinumab 300 mg sc injection every week for 4 weeks followed by Secukinumab 300 mg every 4 weeks until week 100
  Interventions: Biological: Secukinumab
- Placebo arm 1 (Group 4) (Placebo Comparator): Placebo to Secukinumab sc injection every week for 4 weeks followed by placebo to Secukinumab every 4 weeks until week 16. Non-responders will be switched to Secukinumab either 150 or 300 mg sc injection every four weeks until week 100. Responders at week 16 continued receiving placebo until week 24, then were switched to secukinumab 150 or 300 mg sc injection every 4 weeks until week 100. PLEASE NOTE: Placebo arms 1 and 2 belong to the same placebo group (group 4)
  Beginning at Week 52, for subjects whose signs and symptoms were not fully controlled, and who the investigator believed may improve further with an increase in dose, may have had the secukinumab dose increased to 300mg s.c. every 4 weeks.
  Interventions: Biological: Secukinumab
- Placebo arm 2 (Group 4) (Placebo Comparator): Placebo to Secukinumab sc injection every week for 4 weeks followed by placebo to Secukinumab every 4 weeks until week 16. Non-responders were switched to Secukinumab either 150 or 300 mg sc injection every four weeks until week 100. Responders at week 16 continued receiving placebo until week 24, then were switched to secukinumab 150 or 300 mg sc injection every 4 weeks until week 100. PLEASE NOTE: Placebo arms 1 and 2 belong to the same placebo group (group 4)
  Beginning at Week 52, for subjects whose signs and symptoms were not fully controlled, and who the investigator believed may improve further with an increase in dose, may have had the secukinumab dose increased to 300mg s.c. every 4 weeks.
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: Secukinumab — Anti IL-17a monoclonal antibody
  Other Names: AIN457

SUMMARY:
The purpose of this study was to demonstrate efficacy including effect on inhibition of progression of structural damage, safety and tolerability up to 2 years with primary focus at Week 16 (week 24 for structural damage), to support the use of secukinumab pre-filled syringe (PFS) by subcutaneous (s.c.) self-administration with or without loading regimen in subjects with active Psoriatic Arthritis (PsA) despite current or previous NSAID, DMARD therapy and/or previous anti-TNFα therapy. Long term efficacy up to 2 years was based on signs and symptoms of joint/bone structure preservation (X-ray) and improvement in physical function measured by Health Assessment Questionnaire - Disability Index (HAQ-DI©), as well as skin and nail improvement for psoriasis signs.

DETAILED DESCRIPTION:
This multicenter study uses a randomized, double-blind, placebo-controlled, parallel-group design. A screening period (SCR) running up to 10 weeks before randomization will be used to assess subject eligibility followed by 104 weeks of treatment.

At BSL approximately 990 subjects whose eligibility is confirmed will be randomized to one of four treatment groups in 2:2:2:3 ratio:

* Group 1 - secukinumab 150 mg s.c. without loading regimen
* Group 2 - secukinumab 150 mg s.c. with loading dose regimen
* Group 3 - secukinumab 300 mg s.c. with loading dose regimen
* Group 4 - Placebo s.c. NOTE: Group 4 is split into 2 treatment arms, detailed description below. At randomization, subjects will be stratified on the basis of previous anti-TNF therapy as TNFα inhibitor naïve (TNF-naïve) or TNFα inhibitor inadequate responders (TNF-IR).

At each study treatment visit, one (for secukinumab 150 mg) or two (for secukinumab 300 mg) s.c. injections in the form of PFS will be administered, since secukinumab is available in 1.0 mL (150 mg) PFSs. Placebo to secukinumab is also available in 1.0 mL to match the active drug.

At Week 16, subjects who have been randomized to secukinumab groups at BSL (Groups 1-3) will be classified as either responders (≥20% improvement from BSL in both tender joint count (TJC) and swollen joint counts (SJC)) or non-responders (<20% improvement from BSL TJC or SJC), however they will continue on the same treatment irrespective of their response status.

At Week 16, subjects who have been randomized to placebo at BSL (Group 4) will be classified as either responders (≥20% improvement from BSL in both TJC and SJC) or non-responders (<20% improvement from BSL TJC or SJC):

* Subjects who are non-responders will receive either secukinumab 150 mg or 300 mg s.c. every 4 weeks starting at Week 16 (as dictated by treatment sequence assigned to these subjects at BSL).
* Subjects who are responders will continue to receive placebo every 4 weeks. Starting Week 24, these subjects will receive either secukinumab 150 mg s.c. or 300 mg s.c. every 4 weeks starting at Week 24 (as dictated by treatment sequence assigned to these subjects at BSL).

At Week 24, the assessments to address the primary objective will be performed. As described above, subjects who are still receiving placebo s.c. injection will receive either secukinumab 150 mg s.c. or 300 mg s.c. every 4 weeks starting at Week 24 (as dictated by treatment sequence assigned to these subjects at BSL).

At week 52, based on Investigator's decision, the subjects on a 150 mg dose whose signs and symptoms do not show satisfactory response have the possibility to be allocated to secukinumab 300 mg s.c.

After the Week 52 database lock and analyses have been completed, site personnel and subjects will be unblinded to the original randomized treatment (sequence) assignment at randomization. In addition, treatment will be given open-label in order to eliminate the placebo injection. The subject will continue to receive the same active dose of secukinumab as open-label treatment administered until Week 100.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of PsA classified by CASPAR criteria and with symptoms for at least 6 months with moderate to severe PsA who must have at BSL ≥3 tender joints out of 78 and ≥3 swollen joints out of 76 (dactylitis of a digit counts as one joint each).

* Rheumatoid factor (RF) and anti-cyclic citrullinated peptide (anti-CCP) antibodies negative at screening.
* Diagnosis of active plaque psoriasis or nail changes consistent with psoriasis or a documented history of plaque psoriasis.
* Subjects with PsA should have taken NSAIDs for at least 4 weeks prior to randomization with inadequate control of symptoms or at least one dose if stopped due to intolerance to NSAIDs.-Subjects who are regularly taking NSAIDs as part of their PsA therapy are required to be on a stable dose for at least 2 weeks before study randomization and should remain on a stable dose up to Week 24.
* Subjects taking corticosteroids must be on a stable dose of ≤10 mg/day prednisone or equivalent for at least 2 weeks before randomization and should remain on a stable dose up to Week 24.
* Subjects taking MTX (≤ 25 mg/week) are allowed to continue their medication if the dose is stable for at least 4 weeks before randomization and should remain on a stable dose up to Week 52.
* Subjects on MTX must be on folic acid supplementation at randomization.
* Subjects who are on a DMARD other than MTX must discontinue the DMARD 4 weeks prior to randomization visit except for leflunomide, which has to be discontinued for 8 weeks prior to randomization unless a cholestyramine wash-out has been performed.
* Subjects who have been on a TNFα inhibitor must have experienced an inadequate response to previous or current treatment with a TNFα inhibitor given at an approved dose for at least 3 months or have stopped treatment due to safety/tolerability problems after at least one administration of a TNFα inhibitor.
* Subjects who have previously been treated with TNFα inhibitors (investigational or approved) will be allowed entry into study after appropriate wash-out period prior to randomization

Exclusion Criteria:

Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process. - Subjects taking high potency opioid analgesics.

* Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor. - Ongoing use of prohibited psoriasis treatments / medications (e.g., topical corticosteroids, UV therapy) at randomization.
* Any intramuscular or intravenous or intra-articular corticosteroid treatment within 4 weeks before randomization.
* Subjects who have ever received biologic immunomodulating agents except for those targeting TNFα (investigational or approved).
* Previous treatment with any cell-depleting therapies including but not limited to anti- CD20, investigational agents
* Other protocol-defined exclusion criteria do apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (149):
- United States (19):
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Wexford, Pennsylvania
  - Novartis Investigative Site, Wyomissing, Pennsylvania
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, San Miguel de Tucumán
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Canada (6):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Chile (2):
  - Novartis Investigative Site, Vitacura, Santiago Metropolitan
  - Novartis Investigative Site, Santiago
- Czechia (4):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště
- Novartis Investigative Site, Odense, Denmark
- Novartis Investigative Site, Tartu, Estonia
- Novartis Investigative Site, Hyvinkää, Finland
- Germany (11):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Abbach
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Nienburg
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Veszprém
- India (6):
  - Novartis Investigative Site, Secunderabad, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Dublin, Ireland
- Israel (6):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Potenza, PZ
  - Novartis Investigative Site, Udine, UD
- Latvia (4):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Liepāja
  - Novartis Investigative Site, Riga
  - Novartis Investigative Site, Valmiera
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Vilnius
- Mexico (5):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Metepec, State of Mexico
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (4):
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Schiedam
  - Novartis Investigative Site, Utrecht
- Philippines (3):
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Russia (11):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Spain (12):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- Thailand (5):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (19):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Christchurch, Dorset
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Inverness, Invernesshire
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Eastbourne
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Wigan
- Vietnam (3):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Mease P, van der Heijde D, Landewe R, Mpofu S, Rahman P, Tahir H, Singhal A, Boettcher E, Navarra S, Meiser K, Readie A, Pricop L, Abrams K. Secukinumab improves active psoriatic arthritis symptoms and inhibits radiographic progression: primary results from the randomised, double-blind, phase III FUTURE 5 study. Ann Rheum Dis. 2018 Jun;77(6):890-897. doi: 10.1136/annrheumdis-2017-212687. Epub 2018 Mar 17. PMID 29550766
- [Derived] Mease PJ, Coates LC, Gaillez C, Shew A, Bao W, Ritchlin CT. Relationship of radiographic progression status to low disease activity in patients with psoriatic arthritis receiving secukinumab treatment for two years. Rheumatology (Oxford). 2025 Sep 18:keaf488. doi: 10.1093/rheumatology/keaf488. Online ahead of print. PMID 40973471
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Secukinumab in Patients with Psoriatic Arthritis at 52 Weeks Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):817-828. doi: 10.1007/s40744-024-00652-7. Epub 2024 Mar 6. PMID 38446397
- [Derived] Pournara E, Kormaksson M, Nash P, Ritchlin CT, Kirkham BW, Ligozio G, Pricop L, Ogdie A, Coates LC, Schett G, McInnes IB. Clinically relevant patient clusters identified by machine learning from the clinical development programme of secukinumab in psoriatic arthritis. RMD Open. 2021 Nov;7(3):e001845. doi: 10.1136/rmdopen-2021-001845. PMID 34795065
- [Derived] Mease PJ, Landewe R, Rahman P, Tahir H, Singhal A, Boettcher E, Navarra S, Readie A, Mpofu S, Delicha EM, Pricop L, van der Heijde D. Secukinumab provides sustained improvement in signs and symptoms and low radiographic progression in patients with psoriatic arthritis: 2-year (end-of-study) results from the FUTURE 5 study. RMD Open. 2021 Jul;7(2):e001600. doi: 10.1136/rmdopen-2021-001600. PMID 34330846
- [Derived] van der Heijde D, Mease PJ, Landewe RBM, Rahman P, Tahir H, Singhal A, Boettcher E, Navarra S, Zhu X, Ligozio G, Readie A, Mpofu S, Pricop L. Secukinumab provides sustained low rates of radiographic progression in psoriatic arthritis: 52-week results from a phase 3 study, FUTURE 5. Rheumatology (Oxford). 2020 Jun 1;59(6):1325-1334. doi: 10.1093/rheumatology/kez420. PMID 31586420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 173 centers in 28 countries.
Pre-assignment Details: 996 were randomized and dosed, of which 932 participants completed 24 weeks of treatment. Out of the 64 participants who discontinued the most common reasons were participant/guardian decision (32) and adverse events (16).
Groups:
- Secukinumab 150 mg Without Load: Participants were subcutaneously (s.c.) administered with 150 milligrams (mg) of secukinumab as 1 milliliter (mL) Pre-Filled Syringe (PFS) and secukinumab matching placebo (1 mL PFS) at baseline. Participants received secukinumab matching placebo (2*1 mL PFS) at Weeks 1, 2 and 3. From week 4 participants received secukinumab 150 mg (1 mL PFS) and secukinumab matching placebo (1 mL PFS) every four weeks up to 100 weeks.
- Secukinumab 150 mg With Load: Participants were s.c. administered with 150 mg of secukinumab as 1 mL PFS and secukinumab matching placebo (1 mL PFS) at baseline, weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4 up to 100.
- Secukinumab 300 mg With Load: Participants were s.c. administered with 300 mg of secukinumab as 2*1 mL PFS (150 mg dose) at baseline, weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4 up to 100 weeks.
- Placebo: Participants were s.c. administered with secukinumab matching placebo (2*1 mL PFS) at baseline, weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4. Participants were further randomized to two different treatment sequences in 1:1 ratio at baseline as secukinumab matching placebo till Week 16/24 followed by secukinumab 150 mg every 4 weeks starting at Week 16/24 up to 100 weeks and secukinumab matching placebo till Week 16/24 followed by secukinumab 300 mg every 4 weeks starting at Week 16/24 up to 100 weeks.
Period: Overall Study
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Started | 222 | 220 | 222 | 332
Completed (Completed Randomisation phase (up to week 24).) | 207 | 214 | 216 | 295
Not Completed | 15 | 6 | 6 | 37
Not completed — Adverse Event | 2 | 2 | 3 | 9
Not completed — Lack of Efficacy | 3 | 1 | 0 | 3
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 3 | 3 | 19
Not completed — Due to Non-compliance with treatment | 0 | 0 | 0 | 1
Not completed — Due to Technical problems | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomized set was defined as all participants who were randomized.
Groups:
- Secukinumab 150 mg Without Load: Participants were s.c. administered with 150 milligrams (mg) of secukinumab as 1 mL PFS and secukinumab matching placebo (1 mL PFS) at baseline. Participants received secukinumab matching placebo (2*1 mL PFS) at Weeks 1, 2 and 3. From week 4 participants received secukinumab 150 mg (1 mL PFS) and secukinumab matching placebo (1 mL PFS) every four weeks up to 100 weeks.
- Total: Total of all reporting groups
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo | Total
Number analyzed (Participants) | 222 | 220 | 222 | 332 | 996
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.82) | 48.4 (12.87) | 48.9 (12.80) | 49.0 (12.12) | 48.8 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 109 | 114 | 171 | 496
  Male | 120 | 111 | 108 | 161 | 500
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 30 | 31 | 51 | 137
  Not Hispanic or Latino | 180 | 160 | 174 | 251 | 765
  Unknown or Not Reported | 17 | 30 | 17 | 30 | 94
Subjects with psoriasis of hands and feet [Count of Participants; unit: Participants]
  Yes | 133 | 135 | 127 | 174 | 569
  No | 89 | 85 | 95 | 158 | 427
Subjects with psoriasis of nail [Count of Participants; unit: Participants]
  Yes | 153 | 135 | 144 | 231 | 663
  No | 69 | 85 | 78 | 101 | 333
Subjects with psoriasis ≥ 3% of BSA [Count of Participants; unit: Participants]
  Yes | 117 | 125 | 110 | 162 | 514
  No | 105 | 95 | 112 | 170 | 482

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Active Psoriatic Arthritis (PsA) Achieving an American College of Rheumatology Response 20 (ACR20) at Week 16
Description: ACR20 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20% improvement based on tender 78-joint count, swollen 76-joint count and at least 20% improvement in 3 of the following 5 measures: participant's assessment of PsA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, participant's self-assessed disability (Health Assessment Questionnaire Disability Index (HAQ-DI) score), and acute phase reactant evaluated as (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR)).
Time Frame: Week 16
Population: The analysis was performed in Full Analysis Set (FAS) population defined as all randomized participants assigned to study treatment. Following the intent-to-treat principle, participants were analyzed according to treatment assigned at randomization by actual anti-Tumor Necrosis Factor (TNF) status. Missing responses were imputed as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 222 | 220 | 222 | 332
percentage of participants | 59.5 | 55.5 | 62.6 | 27.4
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load vs Placebo; Statistical values were calculated from a logistic regression model with treatment and randomization stratum (TNF-a status -naive or Incidence Rate) as factors and baseline weight as a covariate; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.02, 95% CI 2-sided [2.78 to 5.79]
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.38, 95% CI 2-sided [2.35 to 4.87]
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.58, 95% CI 2-sided [3.16 to 6.63]

2. Secondary Outcome: Change From Baseline to Week 24 With Secukinumab Compared With Placebo for Joint/Bone Structural Damage (Using Van Der Heijde Modified Total Sharp Score (mTSS))
Description: PsA modified vdH-mTSS scoring method was used to assess bone erosion & joint space narrowing (JSN) in hands & feet; that included the 2nd through 5th distal interphalangeal (DIP) joints of each hand. Maximum score for erosions was 5 in joints of the hands and 10 in joints of the feet with 0=no erosions, 1=discrete erosion, 2=large erosion not passing the mid-line, and 3=large erosion passing the mid-line. JSN is: 0=normal, 1=asymmetrical or minimal narrowing up to a maximum of 25%, 2 = definite narrowing with loss of up to 50% of the normal space, 3 = definite narrowing with loss of 50-99% of the normal space, and 4 = absence of a joint space. Maximum erosion score is 320 (200 for the hands and 120 for the feet), and the max total JSN score is 208 (160 for the hands and 48 for the feet). Total radiographic score (hands & feet combined) ranges from 0 to 528, where higher scores indicate more articular damage
Time Frame: Baseline, Week 24
Population: The analysis was performed in FAS population with a measurement that could be evaluated. Participants in placebo group, rescued at Week 16 were also extrapolated (i.e. treated as missing at Week 24).
Measure: Mean (Standard Deviation); unit: Mean Sharp Score
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 222 | 220 | 222 | 332
Mean Sharp Score
  baseline: number analyzed (Participants) | 210 | 213 | 217 | 296
  baseline | 15.25 (37.098) | 13.50 (25.636) | 12.90 (23.781) | 14.95 (38.236)
  change: number analyzed (Participants) | 210 | 213 | 217 | 296
  change | -0.10 (2.872) | 0.13 (1.222) | 0.02 (1.336) | 0.50 (1.708)
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load vs Placebo; Secukinumab 300 mg With Load compared to Placebo Estimate (for the difference in mean), SE and p-value are from a non-parametric ANCOVA model (Koch, 1998) with the change from baseline van der Heijde total modified Sharp score (or Erosion Score or Joint Space Narrowing Score) as the dependent variable, treatment and randomization stratum (TNFa status -naive or IR ) as factors, and weight and baseline van der Heijde total modified Sharp score as covariates; Test type: Superiority; p = 0.0061, Non-parametric ANCOVA model; Difference in Mean = -0.61, Standard Error of Mean 0.22 — *For the Statistical Test of the Hypothesis for the Secondary Outcome, The Estimation Parameter is the Standard Error of the Difference in Mean and not Standard Error of the Mean
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0048, Non-parametric ANCOVA model; Difference in Mean = -0.36, Standard Error of Mean 0.13 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0003, Non-parametric ANCOVA model; Difference in Mean = -0.48, Standard Error of Mean 0.13 — For the Statistical Test of the Hypothesis for the Secondary Outcome, The Estimation Parameter is the Standard Error of the Difference in Mean and not Standard Error of the Mean

3. Secondary Outcome: Count and Percentage of Patients Achieving Psoriatic Area and Severity Index 75 (PASI75) Response
Description: The efficacy of secukinumab 150 mg (with or without loading regimen), or 300 mg (with loading regimen) at Week 16 compared with placebo based on the proportion of patients achieving Psoriatic Area and Severity Index 75 (PASI75) response.
Time Frame: Week 16
Population: Psoriasis subset: The psoriasis subset included all FAS patients who had ≥ 3% of the BSA affected by psoriatic skin involvement at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 117 | 125 | 110 | 162
Participants | 68 | 75 | 77 | 20
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load; Odds ratio, 95% confidence interval, and p-value are from a logistic regression model with treatment and randomization stratum (TNF-alpha status -naïve or IR) as factors and baseline weight as a covariate; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 10.15, 95% CI 2-sided [5.52 to 18.63]
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 11.66, 95% CI 2-sided [6.37 to 21.37]
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 18.06, 95% CI 2-sided [9.56 to 34.12]

4. Secondary Outcome: Count and Percentage of Patients Achieving Psoriatic Area and Severity Index 90 (PASI90) Response
Description: The efficacy of secukinumab 150 mg (with or without loading regimen), or 300 mg (with loading regimen) at Week 16 compared with placebo based on the proportion of patients achieving Psoriatic Area and Severity Index 90 (PASI90) response.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 117 | 125 | 110 | 162
Participants | 37 | 46 | 59 | 15
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load; Odds ratio, 95% confidence interval, and p-value are from a logistic regression model with treatment and randomization stratum (TNF-alpha status -naïve or IR) as factors and baseline weight as a covariate. Missing responses are imputed as non-responders; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.51, 95% CI 2-sided [2.31 to 8.83]
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 6.14, 95% CI 2-sided [3.18 to 11.87]
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 12.55, 95% CI 2-sided [6.43 to 24.48]

5. Secondary Outcome: Count and Percentage of Patients Achieving an ACR50 Response
Description: ACR 50 Response is a measure based on American College of Rheumatology criteria of at least a 50% improvement in the number of tender and swollen joints, and a 50% improvement in at least 3 of the following: the patient's global assessment of disease status; the patient's assessment of pain; the patient's assessment of function measured using the Stanford Health Assessment Questionnaire the physician's global assessment of disease status; serum C-reactive protein levels.
Time Frame: 16 weeks
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 222 | 220 | 222 | 332
Participants | 71 | 79 | 88 | 27
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio, log = 5.37, 95% CI 2-sided [3.30 to 8.73]
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 6.37, 95% CI 2-sided [3.93 to 10.32]
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 7.43, 95% CI 2-sided [4.61 to 12.00]

6. Secondary Outcome: Change From Baseline in HAQ-DI© Score
Description: The change (within treatment) on secukinumab 150 mg (with or without loading regimen), or 300 mg (with loading regimen), at Week 16 compared with placebo for the disease activity assessed by the changes in The Health Assessment Questionnaire disability index (HAQ-DI) relative to baseline.
Time Frame: 16 weeks
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 211 | 210 | 211 | 300
scores on a scale | -0.45 (0.035) | -0.44 (0.035) | -0.55 (0.035) | -0.21 (0.029)
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load; Test type: Superiority — Mixed model with treatment regimen, analysis visit and randomization stratum (TNF-alpha status -naïve or IR) as factors, weight and baseline score as continuous covariates, and treatment by analysis visit and baseline score by analysis visit as interaction terms, using an unstructured covariance structure; p < 0.0001, Mixed Models Analysis; LS Mean, 95% confidence interval, and p-value are from a mixed model for repeated measures (MMRM); Treatment contrast in LS mean (Change) = -0.24, 95% CI 2-sided [-0.32 to -0.15], Standard Error of Mean 0.045
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean, 95% confidence interval, and p-value are from a mixed model for repeated measures (MMRM); Treatment Contrast in LS mean (Change) = -0.23, 95% CI 2-sided [-0.32 to -0.14], Standard Error of Mean 0.045
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean, 95% confidence interval, and p-value are from a mixed model for repeated measures (MMRM); Treatment Contrast inj LS mean (Change) = -0.33, 95% CI 2-sided [-0.42 to -0.24], Standard Error of Mean 0.045

7. Secondary Outcome: Change From Baseline in Disease Activity Score for 28 Joints (DAS28-CRP) (Utilizing High Sensitivity C-Reactive Protein (hsCRP))
Description: The improvement on secukinumab 150 mg (with or without loading regimen), or 300 mg (with loading regimen) at Week 16 compared with placebo for the disease activity assessed by the changes in Disease Activity Score for 28 joints (DAS28-CRP) (utilizing High sensitivity C-Reactive Protein (hsCRP)) relative to baseline.
  Scores range from 0 (no difficulty) to 3 (unable to do)
Time Frame: 16 weeks
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 210 | 208 | 209 | 297
scores on a scale | -1.29 (0.074) | -1.29 (0.075) | -1.49 (0.074) | -0.63 (0.062)
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load; Mixed model with treatment regimen, analysis visit and randomization stratum (TNF-alpha status -naïve or IR) as factors, weight and baseline score as continuous covariates, and treatment by analysis visit and baseline score by analysis visit as interaction terms, using an unstructured covariance structure; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean, 95% CI, and p-value are from a mixed model repeated measures (MMRM); Treatment contrast in LS mean (Change) = -0.66, 95% CI 2-sided [-0.85 to -0.47], Standard Error of Mean 0.096
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean, 95% CI, and p-value are from a mixed model repeated measures (MMRM); Treatment Contrast in LS Mean (Change) = -0.66, 95% CI 2-sided [-0.85 to -0.47], Standard Error of Mean 0.096
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean, 95% CI, and p-value are from a mixed model repeated measures (MMRM); Treatment contrast in LS mean (Change) = -0.86, 95% CI 2-sided [-1.05 to -0.67], Standard Error of Mean 0.096

8. Secondary Outcome: Count and Percentage of Patients With Enthesitis in the Subset of Patients Who Had Enthesitis at Baseline
Description: The efficacy of secukinumab pooled regimen (150 mg with or without loading regimen, and 300 mg with loading regimen) at Week 16 compared with placebo based on the proportion of patients with enthesitis in the subset of patients who had enthesitis at baseline
Time Frame: 16 weeks
Population: Enthesitis subset: The enthesitis subset included all FAS patients who had enthesitis at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 129 | 141 | 140 | 192
Participants | 75 | 64 | 62 | 124
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load; Test type: Superiority; p = 0.2250, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.47 to 1.19]
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.29 to 0.70]
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio, log = 0.44, 95% CI 2-sided [0.28 to 0.69]

9. Secondary Outcome: Count and Percentage of Participants With Dactylitis in the Subset of Patients Who Have Dactylitis at Baseline
Description: The efficacy of secukinumab pooled regimen (150 mg with or without loading regimen, and 300 mg with loading regimen) at Week 16 compared with placebo based on the proportion of patients with dactylitis in the subset of patients who have dactylitis at baseline
Time Frame: 16 weeks
Population: Dactylitis subset: The dactylitis subset included all FAS patients who had dactylitis at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Placebo
Number analyzed (Participants) | 103 | 80 | 82 | 124
Participants | 45 | 34 | 28 | 84
Statistical Analysis 1: Comparison: Secukinumab 150 mg Without Load; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.22 to 0.65]
Statistical Analysis 2: Comparison: Secukinumab 150 mg With Load; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.19 to 0.60]
Statistical Analysis 3: Comparison: Secukinumab 300 mg With Load; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.13 to 0.44]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 24 weeks All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 24 weeks
Description: An Adverse Event (AE) is any sign or symptom that occurs during the study treatment plus 28 days post treatment
Groups:
- Secukinumab 150 mg Without Load: Participants were s.c. administered with 150 milligrams (mg) of secukinumab as 1 mL PFS and secukinumab matching placebo (1.0 mL PFS) at baseline. Participants received secukinumab matching placebo (2*1 mL PFS) at Weeks 1, 2 and 3. From week 4 participants received secukinumab 150 mg (1 mL PFS) and secukinumab matching placebo (1 mL PFS) every four weeks up to 100 weeks.
- Secukinumab 150 mg With Load: Participants were s.c. administered with 150 mg of secukinumab as 1 mL PFS and secukinumab matching placebo (1.0 mL PFS) at baseline, weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4 up to 100.
- Secukinumab Total: Participants were s.c. administered with secukinumab and secukinumab matching placebo at baseline, weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4 up to 100.
Arm/Group | Secukinumab 150 mg Without Load | Secukinumab 150 mg With Load | Secukinumab 300 mg With Load | Secukinumab Total | Placebo
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/220 | 0/222 | 0/822 | 0/332
Serious Adverse Events (participants affected / at risk) | 6/222 | 9/220 | 7/222 | 25/822 | 12/332
Other Adverse Events (participants affected / at risk) | 95/222 | 82/220 | 83/222 | 275/822 | 127/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg Without Load (N=222) | Secukinumab 150 mg With Load (N=220) | Secukinumab 300 mg With Load (N=222) | Secukinumab Total (N=822) | Placebo (N=332)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Typhoid fever (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Computerised tomogram thorax abnormal (Investigations) | 0 | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg Without Load (N=222) | Secukinumab 150 mg With Load (N=220) | Secukinumab 300 mg With Load (N=222) | Secukinumab Total (N=822) | Placebo (N=332)
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 6 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 9 | 21 | 22
Nausea (Gastrointestinal disorders) | 7 | 4 | 3 | 14 | 12
Vomiting (Gastrointestinal disorders) | 3 | 6 | 2 | 12 | 2
Fatigue (General disorders) | 4 | 4 | 4 | 12 | 8
Bronchitis (Infections and infestations) | 3 | 1 | 8 | 12 | 2
Influenza (Infections and infestations) | 2 | 4 | 5 | 12 | 3
Oral herpes (Infections and infestations) | 3 | 0 | 5 | 8 | 4
Rhinitis (Infections and infestations) | 2 | 2 | 7 | 11 | 3
Upper respiratory tract infection (Infections and infestations) | 14 | 17 | 7 | 38 | 11
Urinary tract infection (Infections and infestations) | 6 | 8 | 6 | 20 | 8
Viral upper respiratory tract infection (Infections and infestations) | 13 | 15 | 14 | 44 | 29
Contusion (Injury, poisoning and procedural complications) | 3 | 5 | 2 | 10 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 1 | 0 | 6 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 4 | 8 | 23 | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 | 9 | 3 | 20 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 5 | 3 | 9 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 12 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4 | 4 | 16 | 12
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 7 | 7
Headache (Nervous system disorders) | 8 | 9 | 5 | 23 | 13
Anxiety (Psychiatric disorders) | 1 | 5 | 0 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 4 | 14 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 5 | 16 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 11 | 3 | 16 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 11 | 12
Hypertension (Vascular disorders) | 9 | 5 | 8 | 22 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02404350/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02404350/SAP_001.pdf